CLINICAL TRIAL: NCT01319981
Title: Hyper-CVAD With Liposomal Vincristine (Hyper-CMAD) in Acute Lymphoblastic Leukemia
Brief Title: Hyper-CVAD With Liposomal Vincristine in Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0598; NCI-2011-00861 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; Lymphoblastic lymphoma; Cytoxan; Neosar; Mesnex; Liposomal Vincristine; Vincristine Sulfate Liposomes Injection; Marqibo; Dexamethasone; Adriamycin; Rubex; Cytarabine; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Imatinib Mesylate; Gleevec; ST1571; NSC-716051; Filgrastim; Neupogen
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Rituximab; Imatinib Mesylate; Cyclophosphamide; Doxorubicin; Mesna; Vincristine; Methylprednisolone Hemisuccinate; Methylprednisolone; Methylprednisolone Acetate; Methotrexate; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyper-CMAD + Rituximab (Experimental): Odd Courses 1, 3, 5, 7: Rituximab 375 mg/m2 IV Day 1 & 8 Courses 1 & 3; Imatinib oral 600 mg days 1-14 Course 1 then continuously; Cyclophosphamide 300 mg/m2 IV every; 12 hours for 6 doses; Mesna 600 mg/m2/day IV Days 1-3; Doxorubicin 50 mg/m2 IV CVC Day 4; VSLI 2.25 mg/M2 IV Day 1 & 8; Pegfilgrastim 6 mg/kg after chemotherapy + G-CSF 10 µg/kg/day; Dexamethasone 40 mg IV or P.O. daily days 1-4 and days 11-14 +/- 3 days.
  Interventions: Drug: Rituximab; Drug: Imatinib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Mesna; Drug: VSLI; Drug: G-CSF; Drug: Pegfilgrastim; Drug: Dexamethasone
- Hyper-CMAD (Experimental): Courses 2, 4, 6, 8: Rituximab 375 mg/m2 IV Day 1 & 8 Courses 2 & 4; Imatinib oral 600 mg; Methotrexate 200 mg/m2 IV over 2 hours followed by 8-0- mg/m2 over 22 hours on Day 1; Solu-Medrol 40 mg IV hours approximately every 12 hours +/- 2 hours for 6 doses days 1-3 +/- 3 days; Decadron 40 mg IV or orally 4 times Days 1-4; Ara-C 3 gm/m2 IV every 2 hours, 4 doses on Days 2-3; Pegfilgrastim 6 mg/kg after chemotherapy + G-CSF 10 mg/kg/day.
  Interventions: Drug: Rituximab; Drug: Imatinib; Drug: VSLI; Drug: Solu-Medrol; Drug: Methotrexate; Drug: Ara-C; Drug: G-CSF; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Rituximab — In CD20-positive patients, 375 mg/m2 by vein on day 1 and 8 for Courses 1 and 3; and day 1 and 8 of Courses 2 and 4.
  Other Names: Rituxan
Drug: Imatinib — 600 mg by mouth daily days 1-14 for course 1 and continuously on all other courses for patients who are Philadelphia chromosome positive (Ph+).
  Other Names: Imatinib Mesylate; Gleevec; ST1571; NSC-716051
Drug: Cyclophosphamide — 300 mg/m2 by vein over 3 hours every 12 hours x 6 doses days 1, 2, 3 (total dose 1800 mg/m2) for courses 1, 3, 5, 7
  Other Names: Cytoxan; Neosar
  Arms: Hyper-CMAD + Rituximab
Drug: Doxorubicin — 50 mg/m2 by vein over 24 hours on day 4 after last dose of Cyclophosphamide for courses 1, 3, 5, 7
  Other Names: Adriamycin; Rubex
  Arms: Hyper-CMAD + Rituximab
Drug: Mesna — 600 mg/m2 by vein continuous infusion daily for 24 hours days 1-3 for courses 1, 3, 5, 7
  Other Names: Mesnex
  Arms: Hyper-CMAD + Rituximab
Drug: VSLI — 2.0 mg/m2 by vein on day 1 and day 8 for courses 1, 3, 5, 7
  Other Names: Liposomal Vincristine; Vincristine Sulfate Liposomes Injection; Marqibo
Drug: Solu-Medrol — 40 mg by vein every 12 hours for 6 doses days 1-3 for courses 2, 4, 6, 8.
  Other Names: Methylprednisolone; Depo-Medrol; Medrol
  Arms: Hyper-CMAD
Drug: Methotrexate — 200 mg/m2 IV over 2 hrs followed by 800 mg/m2 over 22 hrs on day 1 beginning after the completion of rituximab for Courses 2, 4, 6, and 8.
  Arms: Hyper-CMAD
Drug: Ara-C — 3 gm/m2 by vein over 2 hours every 12 hours for 4 doses on days 2, 3 for Courses 2, 4, 6, and 8.
  Other Names: Cytarabine; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
  Arms: Hyper-CMAD
Drug: G-CSF — 10 µg/kg/day (rounded) given subcutaneously until neutrophil recovery to 1 x 10^9/L or higher can be substituted or can be added if neutrophils have not recovered to 1 x 10^9/L by day 21.
  Other Names: Filgrastim; Neupogen
Drug: Pegfilgrastim — 6 mg/kg (rounded) within 72 hrs after completion of chemotherapy.
  Other Names: Neulasta
Drug: Dexamethasone — 40 mg by vein or by mouth daily days 1-4 and days 11-14 for courses 1, 3, 5, 7
  Other Names: Decadron
  Arms: Hyper-CMAD + Rituximab

SUMMARY:
Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this clinical research study is to learn if intensive chemotherapy (hyper-CVAD therapy) given in combination with liposomal vincristine (Marqibo), in addition to rituximab for patients who are CD20 positive and/or imatinib, dasatinib, or ruxolitinib for patients with the Philadelphia (Ph) chromosome, can help to control ALL or lymphoblastic lymphoma. The safety of this treatment will also be studied. CD20 is a protein "marker" that is found in leukemia or lymphoma cells.

This is an investigational study. Liposomal vincristine is FDA approved for the treatment of patients with CLL who have relapsed at least 2 times. All of the other study drugs used in this study are FDA approved and commercially available. The combination of liposomal vincristine with the other study drugs is also being used in research only.

Up to 65 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
The Study Drugs:

Adriamycin (doxorubicin) is designed to stop the growth of cancer cells, which may cause the cells to die.

Cyclophosphamide is designed to disrupt with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Cytarabine (Ara-C) is designed to insert itself into DNA (the genetic material of cells) of cancer cells and stop the DNA from repairing itself.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body.

Methotrexate is designed to disrupt cells from making and repairing DNA and "copying" themselves.

Vincristine is designed to disrupt the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Liposomal Vincristine (Marqibo) is designed to help vincristine stay in the bloodstream for a longer time, more specifically target tumor tissue, and deliver more of the drug to a tumor site over a longer period of time. This may increase how effective the drug is and lower the risk of possible side effects in healthy, non-tumor tissue.

Rituximab is a monoclonal antibody that is designed to attach to leukemia cells and activate a series of events that may cause the cancer cells to die.

Tyrosine Kinase Inhibitors (TKI--Imatinib, Dasatinib, or Ruxolitinib) Imatinib is a drug designed to block cancer cells from growing and dividing.

Dasatinib and ruxolitinib are designed to block a protein that cancer may need to grow, survive, or spread.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 groups, based on your already performed diagnostic test for a certain protein, called CD20.

* If you test positive for CD20, you will receive hyper-CVAD therapy plus rituximab.
* If you test negative for CD20, you will receive hyper-CVAD therapy only.

In addition, patients with the Philadelphia chromosome (considered Philadelphia-positive or Ph+) will receive imatinib or dasatinib in either group. Patients with Philadelphia chromosome-like disease will receive dasatinib or ruxolitinib. The study doctor will decide which drug these participants will receive.

Study Drug Administration:

Hyper-CVAD therapy is a combination of 7 chemotherapy drugs: the combination of adriamycin (doxorubicin), cyclophosphamide, and liposomal vincristine, alternating with the combination of cytarabine (Ara-C), dexamethasone, methotrexate, and liposomal vincristine. You will receive the 2 different study drug combinations over 21-28 day "courses." You will begin with Course A treatment and alternate with the Course B treatment every other course. You will stay overnight in the hospital for the first 4-5 days of each course.

For Course A of treatment, you will receive cyclophosphamide, liposomal vincristine, doxorubicin, and dexamethasone.

For Course B of treatment, you will receive methotrexate, cytarabine, and liposomal vincristine.

Courses of treatment on this study will continue to alternate or switch between the Course A study drug combination for all odd number courses (3, 5, and 7) and the Course B study drug combination for all even number courses (4, 6, and 8) for a total of up to 8 courses.

While you are on study, all doses of study drug combinations will be given through a central venous catheter (CVC). A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Course 1:

On Days 1, 2, and 3 you will receive cyclophosphamide by vein over about 24 hours, mesna by vein continuously over 24 hours, and liposomal vincristine by vein over 1 hour +/- 30 minutes (Day 1 only). Mesna is given to help prevent blood in the urine, which is sometimes caused by cyclophosphamide.

On Days 2 and 7, methotrexate then cytarabine will be given by intrathecal (IT) infusion directly into your spinal fluid to lower the risk of the disease spreading to the brain.

On Day 4, you will receive doxorubicin by vein over 24 hours.

On Day 5 or 6, G-CSF will be injected under the skin to help with the recovery of bone marrow cells recovery 24 hours after the dose of study drugs.

On Day 8, you will receive liposomal vincristine by vein over 1 hour +/- 30 minutes.

On Days 1-4 and Days 11-14, dexamethasone will be given by mouth with a glass of water or by vein as a short infusion.

CD20 positive patients only will also receive rituximab by vein over 6 hours, on Days 1 and 8, in addition to receiving all study drugs, as described above. If you are CD20 negative, you will not receive rituximab.

Ph+ participants will receive imatinib by mouth with breakfast and a large glass of water (about 8 ounces) or dasatinib by mouth on Days 1-14 during Course 1.

Patients with Philadelphia chromosome-like disease will receive dasatinib 1 time each day or ruxolitinib 2 times each day on Days 1-14 during Course 1.

Course 2:

On Day 1, you will receive methotrexate by vein over 24 hours.

On Days 2 and 3, you will receive cytarabine by vein over 2 hours every 12 hours for a total of 4 doses. You will also be given citrovorum factor (leucovorin) by vein or by mouth to help prevent the possible side effects of methotrexate.

On Day 5 or 6, G-CSF will be injected under the skin to help with bone marrow recovery 24 hours after the dose of study drugs.

On Days 5 and 8, cytarabine then methotrexate will be given by IT infusion to lower the risk of the disease spreading to the brain.

CD20 positive patients only will also receive rituximab by vein over 4 hours, on Days 1 and 8, in addition to receiving all study drugs, as described above. If you are CD20 negative, you will not receive rituximab.

Ph+ participants will receive imatinib by mouth with breakfast and a large glass of water (about 8 ounces) every day during Courses 2-8. Dasatinib will be given by mouth every day during Courses 2-8.

Patients with Philadelphia chromosome-like disease will receive dasatinib 1 time each day or ruxolitinib 2 times each day.

Course 1 Study Visits:

* Blood (about 5 teaspoons each time) will be drawn weekly for routine tests.
* During Week 2 and 3 or 4, a bone marrow aspirate will be performed to check the status of the disease.
* At the end of Course 1, if the study doctor thinks it is needed, a chest X-ray or CT scan will be performed to check the status of the disease.

If the study doctor thinks it is needed, any of these tests may be repeated at any time while you are receiving the study drug combination.

Radiation Treatment:

If you have lymphoblastic lymphoma and you have enlarged lymph glands in the chest, you may receive radiation treatment to the chest after completing 8 courses of therapy and before you begin maintenance therapy. If you are to receive radiation therapy to the chest, the study doctor will discuss this procedure and its known risks with you in more detail, and you will be given a separate consent form to sign.

Maintenance Therapy -- Non-Ph+ Participants

After completing 8 courses of the study drug combinations, you will begin maintenance therapy for a total of 30 months, and will be interrupted by 2 periods of intensive chemotherapy consolidation courses.

Every month during maintenance therapy:

* You will take 6-mercaptopurine every day by mouth.
* You will receive methotrexate by vein or mouth 1 time every week.
* You will receive liposomal vincristine by vein over 1 hour +/- 30 minutes on Day 1.
* You will take dexamethasone by mouth on Days 1-5 each month.

First intensive chemotherapy consolidation courses:

* Six (6) months after you begin maintenance therapy, you will receive two months of intensive chemotherapy courses.
* First, you will receive cyclophosphamide, liposomal vincristine, doxorubicin, and dexamethasone (similar to Course 1) for Month 6 of therapy.
* About one (1) month later, you will receive methotrexate by vein (at a lower dose than given during Course 2) on Day 1 and pegylated asparaginase by vein over about 2 hours on Day 2. You will be given each drug 1 time each week for a total of 4 weeks for Month 7 of therapy.

About eighteen (18) months after you begin maintenance therapy, you will repeat the intensive chemotherapy courses just described.

Maintenance Therapy -- Ph+ Participants and Participants with Ph-like Disease:

After completing 8 courses of the study drug combinations, you will begin maintenance chemotherapy plus TKI (imatinib or dasatinib if you have Ph+ disease; or dasatinib or ruxolitinib if you have Ph-like disease). Maintenance chemotherapy will be given for a total of 24 months, and will be interrupted by 2 periods of intensive chemotherapy courses and the TKI at 6 and 13 months from the start of maintenance. You will continue receiving the TKI every day from that point on, unless intolerable side effects occur.

Every month during maintenance therapy:

* You will take imatinib, dasatinib, or ruxolitinib every day by mouth.
* You will receive liposomal vincristine by vein over 1 hour +/- 30 minutes on Day 1.
* You will take dexamethasone by mouth on Days 1-5 each month.

Intensive chemotherapy consolidation courses:

°At six (6) and eighteen (18) months after you begin maintenance therapy, you will receive two months of intensive chemotherapy courses. You will receive cyclophosphamide, liposomal vincristine, doxorubicin, and dexamethasone with the TKI (similar to Course 1). If the disease is CD20 positive, you may receive rituximab.

Blood Tests:

During maintenance therapy and the intensive consolidation therapy, you will have blood (about 5 teaspoons) drawn every 4 weeks +/- 4 weeks for routine tests.

After intensive chemotherapy consolidation, for as long as you continue to receive maintenance therapy, blood (about 5 teaspoons) will be drawn every 4 weeks +/- 4 weeks, until maintenance therapy is completed:

Additional Tests while on Study:

Every 3-6 months:

* You will have a bone marrow biopsy performed to check the status of the disease.
* If you have mediastinal disease, you will have a chest x-ray or CT scan.

Length of Study:

You will receive up to 8 courses of therapy. If you are not Ph+, you will continue to receive maintenance therapy for up to 30 months. If you are Ph+, you will continue to receive maintenance therapy for up to 24 months, followed by imatinib or dasatinib alone indefinitely. You will be taken off the study if disease gets worse, you experience intolerable side effects, or the study doctor thinks it is in your best interest.

Additional Information:

If you are 60 years or older, you will receive Course 1 chemotherapy in a protective isolation room to decrease the risk of any infection(s) that you may be exposed to while receiving the Course 1 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed previously untreated ALL or lymphoblastic lymphoma >/= 18 years old. Allow urgent administration of cytarabine/hydrea/atra prior to starting treatment on protocol. Allow previous administration of up to one course of Hyper-CVAD and/or FDA approved TKI.
2. Zubrod performance status </= 3.
3. Adequate liver function (bilirubin </= 3.0 mg/dl unless considered due to tumor) and renal function (creatinine </= 3.0 mg/dl, unless considered due to tumor).
4. No active co-existing malignancy with life expectancy less than 12 months due to that malignancy.
5. All men and women of childbearing potential who are participating in the study must agree to use effective forms of birth control throughout the duration of their treatment.
6. Adequate cardiac function as assessed clinically

Exclusion Criteria:

1. Pregnant or lactating women. Women of childbearing potential (WOCB) must have a blood or urine pregnancy test within 7 days prior to administration of the study drug. (WOCB is defined as a woman who has not undergone hysterectomy or bilateral oophorectomy and has not been naturally postmenopausal for at least 24 consecutive months).
2. Active Grade III-IV cardiac failure as defined by the New York Heart Association criteria, uncontrolled angina or MI within 6 months.
3. Patients with medical conditions that compromise their ability to complete the study or confound interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2013 to November 2020
Groups:
- Hyper-CMAD + Rituximab: Odd Courses 1, 3, 5, 7: Rituximab 375 mg/m2 IV Day 1 & 8 Courses 1 & 3; Imatinib oral 600 mg days 1-14 Course 1 then continuously; Cyclophosphamide 300 mg/m2 IV every; 12 hours for 6 doses; Mesna 600 mg/m2/day IV Days 1-3; Doxorubicin 50 mg/m2 IV CVC Day 4; VSLI 2.25 mg/M2 IV Day 1 & 8; Pegfilgrastim 6 mg/kg after chemotherapy + G-CSF 10 µg/kg/day; Dexamethasone 40 mg IV or P.O. daily days 1-4 and days 11-14 +/- 3 days.
  Rituximab: CD20-positive patients, 375 mg/m2 by vein on days 1 and 8 for Courses 1 and 3; and days 1 and 8 of Courses 2 and 4.
  Imatinib: 600 mg by mouth daily days 1-14 for course 1 and continuously on all other courses for patients who are Philadelphia chromosome positive (Ph+).
  Cyclophosphamide: 300 mg/m2 by vein, 3 hours every 12 hours x 6 doses days 1, 2, 3 (total dose 1800 mg/m2) for courses 1, 3, 5, 7
  Doxorubicin: 50 mg/m2 by vein, 24 hours on day 4 after last dose of Cyclophosphamide for courses 1, 3, 5, 7
  Mesna: 600 mg/m2 by vein continuous daily for 24 hours days 1-3 for courses 1, 3, 5, 7
  VSLI: 2.0 mg/m2 by vein on days 1 and 8 for courses 1, 3, 5, 7
  G-CSF: 10 µg/kg/day (rounded) given subcutaneously until neutrophil recovery to 1 x 10^9/L or higher can be substituted or can be added if neutrophils have not recovered to 1 x 10^9/L by day 21.
  Pegfilgrastim: 6 mg/kg (rounded) within 72 hrs after completion of chemotherapy.
  Dexamethasone: 40 mg by vein or by mouth daily days 1-4 and days 11-14 for courses 1, 3, 5, 7
Period: Overall Study
Arm/Group | Hyper-CMAD + Rituximab | Hyper-CMAD
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyper-CMAD + Rituximab | Hyper-CMAD | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 5 | 7 | 12
Age, Continuous [Median (Full Range); unit: years] | 48 [25 to 77] | 61 [40 to 87] | 60 [28 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 14 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Remission at One Year
Description: The complete remission (CR) is the total number of patients who are in CR at one year divided by the total number of patients who received at least one dose of HCVAD with liposomal vincristine. CR was defined as the presence of </=5% blasts in the bone marrow, with >1x10^9/L neutrophils, >100x10^9/L platelets in the perpherial blood, and no extramedullary disease.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hyper-CMAD + Rituximab | Hyper-CMAD
Number analyzed (Participants) | 15 | 16
Participants | 12 | 13

2. Primary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up. Survival will be measured by the estimated median survival computed by Kaplan-Meier (K-M) analysis, which is the time point at which the cumulative survival drops below 50%, if present. If not present then the median Overall Survival is not reached and not available (NA) as there are an insufficient number of participants with events. In either case ranges are provided for observed survival intervals used in the K-M analysis.
Time Frame: Up to 7 years, 8 months
Population: Median not reached due to insufficient number of participants with events.
Measure: Median (Full Range); unit: Months
Arm/Group | Hyper-CMAD + Rituximab | Hyper-CMAD
Number analyzed (Participants) | 15 | 16
Months | NA [0.3 to 92] — Median not reached due to insufficient number of participants with events. | NA [4.4 to 92] — Median not reached due to insufficient number of participants with events.

3. Primary Outcome: Complete Response Duration
Description: The complete remission (CR) is the total number of patients who are in CR at one year divided by the total number of patients who received at least one dose of HCVAD with liposomal vincristine. CR was defined as the presence of </=5% blasts in the bone marrow, with >1x10^9/L neutrophils, >100x10^9/L platelets in the perpherial blood, and no extramedullary disease. Response date to loss of response or last follow up. Remission duration will be measured by the estimated median remission duration computed by Kaplan-Meier (K-M) analysis, which is the time point at which the cumulative remission duration drops below 50%, if present. If not present then median remission duration is not reached and not available (NA) as there are an insufficient number of participants with events. In either case ranges are provided for observed survival intervals used in the K-M analysis..
Time Frame: Up to 7 years, 8 months
Population: Of the 15 participants in the Hyper-CMAD + Rituximab arm, only 14 responded and are evaluable for Complete Remission Duration (CRD).
Measure: Median (Full Range); unit: Months
Arm/Group | Hyper-CMAD + Rituximab | Hyper-CMAD
Number analyzed (Participants) | 14 | 16
Months | NA [6.6 to 92] — Median not reached due to insufficient number of participants. | NA [3.4 to 92] — Median not reached due to insufficient number of participants.

ADVERSE EVENTS:
Time Frame: Up to 7 years
Groups:
- Hyper-CMAD + Rituximab ALL Ph -; Hyper-CMAD + Rituximab ALL Ph +: Odd Courses 1, 3, 5, 7: Rituximab 375 mg/m2 IV Day 1 & 8 Courses 1 & 3; Imatinib oral 600 mg days 1-14 Course 1 then continuously; Cyclophosphamide 300 mg/m2 IV every; 12 hours for 6 doses; Mesna 600 mg/m2/day IV Days 1-3; Doxorubicin 50 mg/m2 IV CVC Day 4; VSLI 2.25 mg/M2 IV Day 1 & 8; Pegfilgrastim 6 mg/kg after chemotherapy + G-CSF 10 µg/kg/day; Dexamethasone 40 mg IV or P.O. daily days 1-4 and days 11-14 +/- 3 days.
  Rituximab: CD20-positive patients, 375 mg/m2 by vein on days 1 and 8 for Courses 1 and 3; and days 1 and 8 of Courses 2 and 4.
  Imatinib: 600 mg by mouth daily days 1-14 for course 1 and continuously on all other courses for patients who are Philadelphia chromosome positive (Ph+).
  Cyclophosphamide: 300 mg/m2 by vein, 3 hours every 12 hours x 6 doses days 1, 2, 3 (total dose 1800 mg/m2) for courses 1, 3, 5, 7
  Doxorubicin: 50 mg/m2 by vein, 24 hours on day 4 after last dose of Cyclophosphamide for courses 1, 3, 5, 7
  Mesna: 600 mg/m2 by vein continuous daily for 24 hours days 1-3 for courses 1, 3, 5, 7
  VSLI: 2.0 mg/m2 by vein on days 1 and 8 for courses 1, 3, 5, 7
  G-CSF: 10 µg/kg/day (rounded) given subcutaneously until neutrophil recovery to 1 x 10^9/L or higher can be substituted or can be added if neutrophils have not recovered to 1 x 10^9/L by day 21.
  Pegfilgrastim: 6 mg/kg (rounded) within 72 hrs after completion of chemotherapy.
  Dexamethasone: 40 mg by vein or by mouth daily days 1-4 and days 11-14 for courses 1, 3, 5, 7
- Hyper-CMAD ALL Ph +; Hyper-CMAD ALL Ph -: Courses 2, 4, 6, 8: Rituximab 375 mg/m2 IV Day 1 & 8 Courses 2 & 4; Imatinib oral 600 mg; Methotrexate 200 mg/m2 IV over 2 hours followed by 8-0- mg/m2 over 22 hours on Day 1; Solu-Medrol 40 mg IV hours approximately every 12 hours +/- 2 hours for 6 doses days 1-3 +/- 3 days; Decadron 40 mg IV or orally 4 times Days 1-4; Ara-C 3 gm/m2 IV every 2 hours, 4 doses on Days 2-3; Pegfilgrastim 6 mg/kg after chemotherapy + G-CSF 10 mg/kg/day.
  Rituximab: In CD20-positive patients, 375 mg/m2 by vein on day 1 and 8 for Courses 1 and 3; and day 1 and 8 of Courses 2 and 4.
  Imatinib: 600 mg by mouth daily days 1-14 for course 1 and continuously on all other courses for patients who are Philadelphia chromosome positive (Ph+).
  VSLI: 2.0 mg/m2 by vein on day 1 and day 8 for courses 1, 3, 5, 7
  Solu-Medrol: 40 mg by vein every 12 hours for 6 doses days 1-3 for courses 2, 4, 6, 8.
  Methotrexate: 200 mg/m2 IV over 2 hrs followed by 800 mg/m2 over 22 hrs on day 1 beginning after the completion of rituximab for Courses 2, 4, 6, and 8.
  Ara-C: 3 gm/m2 by vein over 2 hours every 12 hours for 4 doses on days 2, 3 for Courses 2, 4, 6, and 8.
  G-CSF: 10 µg/kg/day (rounded) given subcutaneously until neutrophil recovery to 1 x 10^9/L or higher can be substituted or can be added if neutrophils have not recovered to 1 x 10^9/L by day 21.
  Pegfilgrastim: 6 mg/kg (rounded) within 72 hrs after completion of chemotherapy.
Arm/Group | Hyper-CMAD + Rituximab ALL Ph - | Hyper-CMAD + Rituximab ALL Ph + | Hyper-CMAD ALL Ph + | Hyper-CMAD ALL Ph -
All-Cause Mortality (participants affected / at risk) | 4/4 | 0/11 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/4 | 6/11 | 6/10 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 7/11 | 7/10 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CMAD + Rituximab ALL Ph - (N=4) | Hyper-CMAD + Rituximab ALL Ph + (N=11) | Hyper-CMAD ALL Ph + (N=10) | Hyper-CMAD ALL Ph - (N=6)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Back Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 3 (6) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestine Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic Event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (6) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyper-CMAD + Rituximab ALL Ph - (N=4) | Hyper-CMAD + Rituximab ALL Ph + (N=11) | Hyper-CMAD ALL Ph + (N=10) | Hyper-CMAD ALL Ph - (N=6)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal Refulx Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Elevated Prothrombin Time (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (2) | 5 (5) | 5 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT01319981/Prot_SAP_ICF_000.pdf